CLINICAL TRIAL: NCT06146621
Title: Targeting Access and Knowledge of Earned Income Tax Credit (EITC) Utilization and Policies
Acronym: TAKE-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: University of California, Berkeley (Other); Boston University (Other); University of California Nutrition Policy Institute (Unknown); University of California, Merced (Other); Blue Shield of California Foundation (Unknown)
Responsible Party: Principal Investigator, Rita Hamad, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA-0221018
Record Dates: First submitted 2023-11-07; First posted 2023-11-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Issue; Food Security; Well-being
Keywords: poverty, safety net

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Information about free tax-filing support (Active Comparator): Basic information about where to find free tax filing support in their community will be provided to all participants by email once upon enrollment.
  Interventions: Behavioral: Information about free tax-filing support
- Low-touch text messaging (Experimental): To address families' lack of awareness of the Earned Income Tax Credit (EITC) and the ways they may benefit from filing taxes, one study arm will receive low-touch text messages. These act in part by increasing awareness of programs and eligibility rules and in part as reminders to overcome limited attention to filing. Study participants receiving this intervention will receive behavioral science-informed text messages in English or Spanish from WIC that inform them about the EITC throughout tax season (i.e., January-April) 2024. We will personalize message contents (e.g., EITC benefit size mentioned in message based on participant income, marital status, and number of dependents) due to suggestive evidence that a tailored, individualized text message has the potential to be effective
  Interventions: Behavioral: Low-touch text messaging; Behavioral: Information about free tax-filing support
- Personal tax filing support (Experimental): Participants randomized to this intervention will be connected with a human assistor who will work with them to ensure they access resources to help them file taxes and apply for the EITC. The English- and Spanish-speaking assistors will be study team staff trained to provide personalized support to help families access resources for which they are eligible. The assistor will be available by text or phone to talk with people if they encounter barriers and will call to follow-up on a mutually agreed upon schedule.
  Interventions: Behavioral: Personal tax filing support; Behavioral: Information about free tax-filing support
- Financial assistance (Experimental): Participants randomized to this intervention will receive a $100 cash incentive for tax filing, designed to offset the time, hassle, and resources spent on tax preparation and filing, as well as psychological frictions like inattention that prevent some people from filing. This will be provided to recipients as soon as they show proof of tax filing, to provide a more immediate reward relative to the delays in receiving a federal tax refund. We will test the feasibility of delivering this via gift card, check, or other modalities, in addition to evaluating the framing and incentive amount.
  Interventions: Behavioral: Information about free tax-filing support; Behavioral: Financial assistance

INTERVENTIONS:
Behavioral: Low-touch text messaging — To address families' lack of awareness of the Earned Income Tax Credit (EITC) and the ways they may benefit from filing taxes, one study arm will receive low-touch text messages. These act in part by increasing awareness of programs and eligibility rules and in part as reminders to overcome limited attention to filing. Study participants receiving this intervention will receive behavioral science-informed text messages in English or Spanish from WIC that inform them about the EITC throughout tax season (i.e., January-April) 2024. We will personalize message contents (e.g., EITC benefit size mentioned in message based on participant income, marital status, and number of dependents) due to suggestive evidence that a tailored, individualized text message has the potential to be effective
  Arms: Low-touch text messaging
Behavioral: Personal tax filing support — Participants randomized to this intervention will be connected with a human assistor who will work with them to ensure they access resources to help them file taxes and apply for the EITC. The English- and Spanish-speaking assistors will be study team staff trained to provide personalized support to help families access resources for which they are eligible. The assistor will be available by text or phone to talk with people if they encounter barriers and will call to follow-up on a mutually agreed upon schedule.
  Arms: Personal tax filing support
Behavioral: Information about free tax-filing support — Basic information about where to find free tax filing support in their community will be provided to all participants by email once upon enrollment.
Behavioral: Financial assistance — Participants randomized to this intervention will receive a $100 cash incentive for tax filing, designed to offset the time, hassle, and resources spent on tax preparation and filing, as well as psychological frictions like inattention that prevent some people from filing. This will be provided to recipients as soon as they show proof of tax filing, to provide a more immediate reward relative to the delays in receiving a federal tax refund. We will test the feasibility of delivering this via gift card, check, or other modalities, in addition to evaluating the framing and incentive amount.
  Other Names: Cash incentive
  Arms: Financial assistance

SUMMARY:
The earned income tax credit (EITC) is the largest United States poverty alleviation program, providing up to $6,600 for working families as a tax refund. Prior studies have shown the EITC's benefits for social outcomes and health. Effects are even more significant for single mothers and Black women. Despite these known benefits, 20%-33% of eligible individuals do not receive benefits, leaving $7 billion unclaimed annually. The Targeting Access and Knowledge of EITC Utilization and Policies (TAKE-UP) Study is a pilot randomized controlled trial that will develop and test the feasibility of several culturally tailored, scalable interventions to increase the take-up of the EITC among participants in the Special Supplemental Food Program for Women, Infants, and Children (WIC).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Special Supplemental Nutrition Program for Woman, Infants, and Children (WIC)
* Eligible for but did not receive the Earned Income Tax Credit (EITC) in the prior tax year
* At least one dependent under 18 years
* Having earned income (including income of spouse, if applicable) for the current tax year within EITC eligibility thresholds based on marital status and number of dependents
* English or Spanish-speaking
* Living in California and not planning to move within the next year
* Immigration status compatible with EITC eligibility
* Access to a phone that receives text messages
* Willing to share relevant fields from tax forms if filing taxes (e.g., adjusted gross income)
* Willing to be randomized.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 84 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who filed taxes | 0-12 months after intervention
  Determine whether participants filed taxes in the 2022 tax year
Number of participants who received the EITC | 0-12 months after intervention
  Determine whether participants received the EITC in the 2022 tax year

SECONDARY OUTCOMES:
Number of participants living with material hardship. Survey instrument: Housing Insecurity/Instability/Homelessness Questions from Social Interventions Research & Evaluation Network (SIREN) at University of California San Fransisco (UCSF) | 0-12 months after intervention
  Evaluate an individual's level of material hardship: whether participant can afford housing, medical care, utilities/if their housing has basic utilities like stove/refrigerator.
Number of participants living with depressive symptoms. Survey Instrument: General Anxiety Disorder-7 | 0-12 months after intervention
  Evaluate an individual's level of depressive symptoms with a 5 point scale for how often depressive symptoms were experienced. Lowest point on scale: none of time, highest point on scale: all of the time. Higher points on scale indicated higher levels of depressive symptoms.
Number of participants living with food insecurity. | 0-12 months after intervention
  6-item United States Department of Agriculture (USDA) food security scale. Lowest point on scale: Never true, Highest Point on scale: Often true. Higher points on scale indicated higher levels of food insecurity.
Number of hours spent tax filing | 0-12 months after intervention
  Amount of hours participant spent tax filing
Number of participants living with anxiety/perceived stress. Survey Instrument: General Anxiety Disorder-7 | 0-12 months after intervention
  Evaluate an individual's level of anxiety/perceived stress with a 5 point scale for how often anxiety/perceived stress was experienced. Lowest point on scale: none of time, highest point on scale: all of the time. Higher points on scale indicated higher levels of anxiety/perceived stress.
Amount of money spent on tax filing | 0-12 months after intervention
  Dollar amount that participant spent on tax filing

CONTACTS AND LOCATIONS:
Overall Officials: Wendi Gosliner, DrPH, Principal Investigator — University of California Nutrition Policy Institute
Locations (1):
- California Special Supplemental Nutrition Program for Women, Infants, and Children (WIC), Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Interested and qualified third-party researchers can apply to access de-identified data used in this study by contacting the PIs.